CLINICAL TRIAL: NCT01363258
Title: Reducing Care-Resistant Behaviors During Oral Hygiene in Persons With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Rita A. Jablonski, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R01NR012737 (NIH)
Record Dates: First submitted 2011-05-27; First posted 2011-06-01 (Estimated); Results first posted 2018-06-07 (Actual); Last update posted 2018-06-07 (Actual); Status verified 2018-05

CONDITIONS: Care-resistant Behavior; Dementia
Keywords: Elderly; Dementia; Care-resistant behavior; Oral health; Long-term care
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Care-resistant mouth care (MOUTh) (Experimental): These nursing home residents with dementia receive mouth care from study personnel who use strategies to reduce care-resistant behavior (Managing Oral Hygiene Using Threat Reduction or MOUTh) while providing evidence-based mouth care.
  Interventions: Behavioral: Care-resistant mouth care (MOUTh)
- Evidence Base Mouth Care (Active Comparator): Nursing home residents with dementia received mouth care from study personnel who were trained in evidence-based mouth care only.
  Interventions: Procedure: Evidence-based mouth care

INTERVENTIONS:
Behavioral: Care-resistant mouth care (MOUTh) — The intervention combines best mouth care practices with a constellation of behavioral techniques that reduce threat perception and thereby prevent or de-escalate care-resistant behavior.
  Arms: Care-resistant mouth care (MOUTh)
Procedure: Evidence-based mouth care — Mouth care tailored to the needs of older adults, including care of dentures.
  Arms: Evidence Base Mouth Care

SUMMARY:
The main purpose of this study is to test a method of providing mouth care to persons with dementia who live in nursing homes. The method of providing mouth care is designed to reduce fear in persons with dementia, so that these persons do not resist mouth care.

DETAILED DESCRIPTION:
Nursing home (NH) residents with dementia are often dependent on others for mouth care, yet will react with care-resistant behavior (CRB) when receiving assistance. The oral health of these elders deteriorates in the absence of daily oral hygiene, predisposing them to harmful systemic problems such as pneumonia, hyperglycemia, cardiac disease, and cerebral vascular accidents. The purpose of this study is to determine whether CRBs can be reduced, and oral health improved, through the application of an intervention based on the neurobiological principles of threat perception and fear response. When faced with a threat, all organisms react with "flight-fight" responses. These responses are both autonomic (e.g. elevated heart rate, sweating) and behavioral (e.g. moving away, attacking). Persons with dementia have heightened threat perception as a result of neurobiological changes that affect the cerebral cortex, hippocampus, and amygdala. These individuals may interpret mouth care as a threatening action by threatening people. The intervention, called Managing Oral Hygiene Using Threat Reduction (MOUTh), combines best mouth care practices with a constellation of behavioral techniques that reduce threat perception and thereby prevent or de-escalate CRB. The primary specific aims of the study are to: 1)Evaluate the efficacy of the MOUTh intervention for reducing CRBs in persons with dementia; 2)Validate the overall efficacy of the MOUTh intervention using nurse-sensitive oral health outcomes--swollen and bleeding gums, cleanliness of the oral cavity, saliva, and integrity of the lips and oral mucosa; and 3)Calculate the cost of the MOUTh intervention. Using a randomized repeated measures design, 80 elders with dementia from 5 different NHs will be randomized at the individual level to the experimental group, which will receive the intervention, or to the control group, which will receive standard mouth care from research team members who receive training in the proper methods for providing mouth care but no training in resistance recognition or prevention/mediation. Oral health assessments and CRB measurements will be obtained during a 7-day observation period and a 21-day intervention period. Individual growth models using multilevel analysis will be used to estimate the efficacy of the intervention for reducing CRBs in persons with dementia, and to estimate the overall efficacy of the intervention using oral health outcomes. Activity-based costing methods will be used to determine the cost of the MOUTh intervention. At the end of this study, the research team anticipates having a proven intervention that prevents and reduces CRB within the context of mouth care. Long-term objectives include testing the effect of the intervention on systemic illnesses among persons with dementia; examining the transferability of this intervention to other activities of daily living; and disseminating threat reduction interventions to NH staff, which may radically change the way care is provided to persons with dementia.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* age 55 or older
* documented diagnosis of dementia, Alzheimer's disease, vascular dementia, or Lewy body dementia
* identified by NH staff as resistant to mouth care
* at least 2 adjacent teeth AND/OR daily wearing of at least one denture plate
* the ability to hold a toothbrush
* the ability to move his or her hand to his or her mouth.

Exclusion Criteria:

* age less than 55
* no documented diagnosis of dementia
* inability to hold a toothbrush
* inability to raise his or her hand to his or her mouth
* receiving treatment for an active dental or denture problem
* a diagnosis of dysphagia requiring thickened liquids

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-04; Primary Completion 2015-08 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rita A Jablonski-Jaudon, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (4):
- United States (4):
  - Centre Crest, Bellefonte, Pennsylvania
  - Spring Creek Rehabilitation &Health Care Center, Harrisburg, Pennsylvania
  - Rest Haven Rehabilitation &Nursing Center, York, Pennsylvania
  - Pleasant Acres Nursing &Rehabilitation Center, York, Pennsylvania

REFERENCES:
- [Background] Jablonski RA, Therrien B, Mahoney EK, Kolanowski A, Gabello M, Brock A. An intervention to reduce care-resistant behavior in persons with dementia during oral hygiene: a pilot study. Spec Care Dentist. 2011 May-Jun;31(3):77-87. doi: 10.1111/j.1754-4505.2011.00190.x. PMID 21592161
- [Derived] Jablonski RA, Kolanowski A, Therrien B, Mahoney EK, Kassab C, Leslie DL. Reducing care-resistant behaviors during oral hygiene in persons with dementia. BMC Oral Health. 2011 Nov 19;11:30. doi: 10.1186/1472-6831-11-30. PMID 22100010

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred sequentially in 9 United States NHs.
Pre-assignment Details: Once potential participants were identified, we obtained consent from the legally authorized representative, screened them against inclusion/exclusion criteria, and then randomly assigned them to control or experimental groups.
Groups:
- Control: Received twice daily standard mouth care for 21 days from research team members. Briefly, all tooth and tongue dorsum surfaces were brushed using a soft toothbrush and fluoride toothpaste. Interdental cleaning was accomplished using interdental brushes. After interdental cleaning, participants rinsed and spit using non-alcoholic antimicrobial (0.07% cetylpyridium chloride) mouth rinse.
- Experimental: The Managing Oral Hygiene Using THreat Reduction (MOUTh) intervention contained 3 components: an evidence-based mouth care protocol for older adults with natural dentition and dentures [all tooth and tongue dorsum surfaces were brushed using a soft toothbrush and fluoride toothpaste. Interdental cleaning was accomplished using interdental brushes. After interdental cleaning, participants rinsed and spit using non-alcoholic antimicrobial (0.07% cetylpyridium chloride) mouth rinse] , recognition of CRBs, and strategies to reduce threat perception during the provision of mouth care.
Period: Overall Study
Arm/Group | Control | Experimental
Started | 54 | 46
Completed | 54 | 46
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Experimental | Total
Number analyzed (Participants) | 54 | 46 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 80.48 (11.54) | 82.80 (8.92) | 81.55 (9.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 31 | 71
  Male | 14 | 15 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 54 | 46 | 100
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 8 | 16
  White | 46 | 38 | 84
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 54 | 46 | 100
Months in nursing home [Mean (Standard Deviation); unit: months] | 17.39 (15.99) | 28.74 (29.16) | 22.66 (23.63)
Global Deterioration Scale [Mean (Standard Deviation); unit: units on a scale] — The Global Deterioration Scales is an ordinal measure that captures the severity of the dementia based on cognitive and functional abilities. Ranges from 1 (normal) to 7 (severe dementia).
  units on a scale | 5.69 (1.03) | 5.73 (0.71) | 5.71 (0.89)
Katz Index of ADLs [Mean (Standard Deviation); unit: units on a scale] — The Katz Index of Activities of Daily Living is an ordinal measure of functional abilities. Higher numbers denote greater impairment, where 0 is completely independent and 18 is completely dependent on others for care.
  units on a scale | 9.33 (2.67) | 9.76 (3.63) | 9.53 (3.16)
Charlson Comorbidity Index [Mean (Standard Deviation); unit: units on a scale] — The Charlson Comorbidity Index assigns weighted values to specific medical conditions, for example, a diagnosis of hypertension may receive a "1" while a diagnosis of uncontrolled diabetes may receive a "2." The higher the number, the more severe the accompanying medical conditions.
  units on a scale | 2.40 (1.53) | 2.60 (2.56) | 2.50 (2.06)

OUTCOME MEASURES:

1. Primary Outcome: Care-Resistant Behavior
Description: Care-resistant behavior will be measured using the Resistiveness to Care Scale.This instrument is a checklist. The 13 care-resistant behaviors (e.g., turn away, hit/kick, say "no", etc.) are listed on the left side of the instrument. There are 3 columns for each behavior (mild, moderate, and severe). When behaviors occur, a tick mark is placed in the appropriate column (mild, moderate, or severe). The final score is obtained by multiplying the sums for mild by 1, the sums for moderate by 2, and the sums for severe behavior by 3. These subtotals are then summed together for a final care-resistant behavior score. One cannot determine the frequency and quality of behaviors from raw scores alone. For example, a score of 12 could mean 12 "mild" behaviors or 4 "severe" behaviors. The sums were used as global care-resistant behavior. Higher numbers signify more frequent and intense care-resistant behavior. Minimum value was 0, max value was 25.
Time Frame: Baseline (observation) to follow-up (week 3)
Population: One-hundred nine NH residents were enrolled; 101 were randomized, 100 contributed data for analyses, and 91 completed the 3-week intervention period.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Control | Experimental
Number analyzed (Participants) | 54 | 46
units on a scale
  Observation (Baseline) | 4.84 (0.66) | 6.3 (0.86)
  Follow-up (Week 3) | 4.42 (0.48) | 4.91 (0.53)
Statistical Analysis 1: Comparison: Control vs Experimental; Test type: Other — Generalized linear mixed models fitted with binomial (logit link) and gamma (log link) distributions, with additional dispersion parameters, were used to estimate and test intervention effects in terms of occurrence and intensity of CRBs, respectively. Inference was conducted in the link scale, but inverse-link estimates in the original scales (proportions and CRB scores, for the binomial and gamma models, respectively) were computed to facilitate interpretation; p = 0.1433, Time by group interaction test; Effect size = -0.16

2. Secondary Outcome: Oral Health
Description: The oral health will be measured as the total score obtained from the Oral Health Assessment Tool. The OHAT contains 8 categories (e.g., status of gums, dentition, moisture of oral cavity, general cleanliness, etc.). Each category is assigned a value of 0=healthy, 1=problematic, and 2=unhealthy. Scores range from 0 (healthy) to 16 (unhealthy).
Time Frame: Baseline (observation) to follow-up (week 3)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Control | Experimental
Number analyzed (Participants) | 54 | 46
units on a scale
  Observation (Baseline) | 4.93 (0.68) | 4.86 (0.68)
  Follow-up (Week 3) | 3.83 (0.62) | 3.42 (0.61)

ADVERSE EVENTS:
Arm/Group | Control | Experimental
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/46
Other Adverse Events (participants affected / at risk) | 0/54 | 0/46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No